CLINICAL TRIAL: NCT04632498
Title: Investigating Biological Markers, Targets, and Intervention for Mood Disorders
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Phase I enrolment and testing completed. Future Phase II enrolment/testing is anticipated.
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, David J. Kennedy, Professor and Chair, Department of Physical Medicine & Rehabilitation, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: IRB #201645
Record Dates: First submitted 2020-10-29; First posted 2020-11-17 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-04

CONDITIONS: Major Depressive Disorder; Depression; Stress
Keywords: EEG/ERP; Neurophysiology; Endocrine; Cognitive; Mindfulness; Mechanistic Clinical Trial
MeSH Terms: conditions — Depressive Disorder, Major; Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mindfulness Based Intervention (MBI) (Experimental): Patients Active Intervention group
  Interventions: Behavioral: Mindfulness Based Intervention
- Wait-list Control (WL) (No Intervention): Patient Control receiving no treatment
- Healthy Control (HC) (No Intervention): Healthy Control receiving no treatment

INTERVENTIONS:
Behavioral: Mindfulness Based Intervention — Standardized 8-week Cognitive and Behavioral Psychotherapy group with 26 hrs of in-class training and homework, along with 1 all-day retreat in which core mindfulness skills are developed
  Other Names: MBI
  Arms: Mindfulness Based Intervention (MBI)

SUMMARY:
This multi-modal methods study will investigate neurophysiological, endocrinological, cognitive, psycho-social-emotional markers of disease, and targets for integrative health treatments in mood disorders.

DETAILED DESCRIPTION:
It is estimated that 16.2 million adults in the USA suffer at least one depressive episode any given year. Mood disorders are associated with decreased quality of life, attention, memory, and executive function deficits, and increased health care cost. Despite successful medication and psychotherapies, mood disorders rarely respond completely to common treatment options. MBI's offer a low-cost, non-pharmacological alternative with accruing efficacy. Developing robust and specific non-pharmacologic intervention programs, on par with pharmacological clinical outcomes without harmful side-effects is a crucial unmet clinical need and a research priority for the NCCIH. Understanding the mechanistic pathways of these interventions is key to their clinical development and implementation for treating depression in primary care.

Mindfulness-Based Interventions (MBIs) show similar clinical efficacy for mood disorders as pharmacology, and co-morbid symptoms of depression and anxiety. There is substantial consistent and replicated empirical evidence across multiple clinical sites highlighting the clinical efficacy of MBI in decreasing risk of depressive relapse ascertained from randomized RCTs comparing MBI with treatment as usual. Meta-analysis including 183 patients with Multiple Sclerosis showed efficacy in psychosocial outcomes, quality of life, anxiety, depression, and select physical symptoms including fatigue, pain, and vestibular symptoms. The clinical efficacy of MBIs appears to extend mood disorders, as a systematic review including 13 studies in fibromyalgia, chronic fatigue, and irritable bowel syndrome showed significant effect sizes, reported as standardized mean difference (SMD), compared to control conditions in reducing depression (SMD= -.23), anxiety (SMD= -.20), symptom severity (SMD= -.40), and pain (SMD= -.21). Cognitively, MBIs appear to enhance executive control and self-regulatory processing, that has a beneficial effect upon emotion regulation, pain perception, and has shown to reduce rumination in depression.

This overarching study aims to identify key phenotypic markers and treatment targets of mood disorders, and further understand MBI mechanism in its treatment.

ELIGIBILITY:
Inclusion Criteria for Patients:

* Age range: 18-65 years
* Must possess English language skills sufficient for providing informed consent, completing questionnaires, and understanding instructions
* If currently taking maintenance anti-depressant and/or anti-anxiety medication, must have a "stable" regimen as indexed by no medication or dosage changes within the past month
* IDS score ≥18
* Currently depressed patients will be defined as: PHQ-9 score range 15 - 27 (moderately severe/severe depressive severity)
* Remitted depressed patients will be defined as: number of depressive episodes must be ≥ 3 and a PHQ-9 score of < 5 (minimal depression)

Blood Collection Inclusion:

* At least 110 pounds
* Generally healthy by self-report on day of collection (i.e., free of cold and flu symptoms on the day of collection, no infections within two weeks prior to collection, no known sickle cell disease)
* Including the study draw, blood donation for clinical or research purposes within the preceding eight weeks will not exceed 550 mL
* No more than one blood draw will have occurred during the preceding week

Exclusion Criteria for Patients:

* Prior diagnosis of bipolar I, bipolar II, psychotic personality disorder, borderline personality disorder, and/or narcissistic personality disorder
* Current history (equal/less than 6 months) of substance abuse/dependence
* Current history (equal/less than 6 months) of regular meditation practice (>1 session/week; >10 min/session)
* History of medical illness associated with possible changes in cerebral tissue or cerebrovasculature (e.g., stroke) or with neurologic abnormality (e.g., seizure disorder, cerebrovascular or neoplastic lesion, neurodegenerative disorder, or significant head trauma, defined by loss of consciousness of ≥ 5 minutes)
* Current suicidal ideation

Exclusion Criteria for Healthy Controls:

* Previous or current mental health history (depression)
* Current history (equal/less than 6 months) of substance abuse/dependence
* History of medical illness associated with possible changes in cerebral tissue or cerebrovasculature (e.g., stroke) or with neurologic abnormality (e.g., seizure disorder, cerebrovascular or neoplastic lesion, neurodegenerative disorder, or significant head trauma, defined by loss of consciousness of ≥ 5 minutes)
* Current suicidal ideation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2021-10-26 (Actual); Primary Completion 2022-01-15 (Actual); Study Completion 2024-04-03 (Actual)

PRIMARY OUTCOMES:
Electroencephalography (EEG) | 36 months
  Event-Related Potentials (ERPs)
Electroencephalography (EEG) | 36 months
  Oscillatory Activity

SECONDARY OUTCOMES:
Endocrine Measures | 36 months
  Oxytocin, Cortisol
Cognitive Behavioral Measure | 36 months
  Executive Functioning
Cognitive Behavioral Measure | 36 months
  Working Memory
Cognitive Behavioral Measure | 36 months
  Social Emotional Processing

OTHER OUTCOMES:
Clinical Measures | 36 months
  Depression Symptoms
Clinical Measures | 36 months
  Anxiety Symptoms
Five Facet Mindfulness Questionnaire (FFMQ) | 36 months
  A 39-item assessment of trait mindfulness (encompassing observing, describing, acting with awareness, non-judging, and non-reactivity).
Rumination Response Scale (RRS) | 36 months
  22-item assessment that reliably assesses rumination and not confounded by depression. The 22 items of the RRS measure two aspects of rumination, brooding and reflective pondering.

CONTACTS AND LOCATIONS:
Overall Officials: Poppy LA Schoenberg, PhD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
The PI will adhere to the NIH Sharing of Biomedical Research Resources: Guidelines for Recipients of NIH Grants and Contracts on Obtaining and Disseminating Biomedical Research Resources.
  1. Quality-controlled raw data as well as processed data used in publications will be de-identified before sharing upon "reasonable request". As described in the proposal, workflows and structure will be exactly described in reports and documented to allow precisely reproduce results from raw data and replicate methodology. Final data (computerized datasets with raw data and derived variables) that have not yet been published will be shared in a timely manner.
  2. Software programs (i.e. experimental paradigm scripts produced for this study) and documentation will be made available for research purposes to replicate findings upon "reasonable request", and any software/script sharing requirements by journals.
Supporting Information: CSR
Time Frame: 36 months